CLINICAL TRIAL: NCT02699749
Title: An Open-Label, Phase 1, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-931, a Cell Division Cycle 7 (CDC7) Inhibitor, in Adult Patients With Advanced Nonhematologic Tumors
Brief Title: A Study to Evaluate TAK-931 in Participants With Advanced Nonhematologic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-931-1002 Merge to Takeda; U1111-1181-0269 (Registry Identifier: WHO); JapicCTI-163200 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-02-29; First posted 2016-03-04 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Nonhematologic Neoplasms, Advanced
Keywords: Drug Therapy
MeSH Terms: interventions — simurosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-931 (Experimental): TAK-931 30 mg, capsules, orally, QD or BID on Days 1-14 of each 21-day treatment cycle in dosing schedule A followed by dosing schedule B, C, D, E and F. In dosing schedules B through F, starting doses and dosing escalations will vary depending on the dosing data obtained from dosing in the previous schedule.
  Dose escalation of TAK-931 will be based on evaluation of clinical safety and tolerability and guided by accumulating PK data. 3-4 dose cohorts are expected for each dosing schedule.
  If the PK from the early cohorts support BID dosing, then study drug administration in subsequent cohorts may transition to a BID dosing schedule.
  Interventions: Drug: TAK-931

INTERVENTIONS:
Drug: TAK-931 — TAK-931 oral capsules.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and maximum tolerated dose (MTD) of TAK-931 in participants with advanced nonhematologic tumors.

DETAILED DESCRIPTION:
The drug being under investigation in this study is called TAK-931. The effect of TAK-931 is being evaluated in up to 100 participants who have nonhematologic (solid) neoplasms. This study will look at the safety, tolerability, and PK to determine the maximum tolerated dose (MTD) of TAK-931.

This multi-center trial will be conducted in Japan. The overall study duration is approximately 42 months for total of dose escalation cohorts and the safety expansion cohort. Participants will make multiple visits to the clinic with final visit approximately 30-40 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of an advanced, nonhematologic/solid tumor (with the exception of primary brain tumor).
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 .
3. For whom no effective standard therapy is available.
4. Life expectancy of greater than or equal to (>=3) months.
5. Female participants who:

   * Are postmenopausal (natural amenorrhea and not due to other medical reasons) for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilized (example, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
   * Agree not to donate sperm during this study and for 120 days after receiving their last dose of study drug.
6. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
7. Ability to swallow oral medications, willingness to undergo serial skin punch biopsies, and suitable venous access for the study-required PK and pharmacodynamic sampling.
8. Clinical laboratory values as specified below within 28 days before the first dose of study drug:

   * Bone marrow reserve consistent with absolute neutrophil count (ANC) >=1500 per millimeter cube (/mm˄3), platelet count >=100,000/mm˄3, and hemoglobin >=9 per gram deciliter (g/dL).
   * Total bilirubin must be less than (<) 1.5 times the upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be 3 <=ULN. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of hepatocellular carcinoma, biliary tract cancer, or metastatic disease in liver.
   * Serum albumin >=3.0 g/dL.
   * Serum creatinine <1.5 times the institutional ULN or creatinine clearance based on the Cockcroft-Gault estimate >=50 milliliter per minute (mL/minute) for participants with serum creatinine concentrations above institutional limits.
9. Left ventricular ejection fraction (LVEF) greater than (>) 50 percent (%) as measured by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 4 weeks before receiving the first dose of study drug.
10. Recovered (that is, <=Grade 1 toxicity) from the reversible effects of prior anticancer therapy. Participants with ongoing toxicities at baseline may be eligible; however, any Grade 2 baseline toxicity (except for alopecia) should be discussed with the medical monitor.

Exclusion Criteria:

1. Who require continuous use of proton pump inhibitors (PPIs) or histamine-2 (H2) receptor antagonists and participants who are taking PPIs within 5 days before the first dose of study drug.
2. Treatment with clinically significant enzyme inducers within 14 days before the first dose of study drug.
3. Treatment with any investigational products within 30 days before the first dose of study drug.
4. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before the first dose of study drug.
5. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
6. History of any of the following within the last 3 months before administration of the first dose of study drug:

   * Ischemic myocardial event including angina requiring therapy and artery revascularization procedures, myocardial infarction, and unstable symptomatic ischemic heart disease.
   * Ischemic cerebrovascular event, including transient ischemic attack and artery revascularization procedures.
   * Thromboembolic events (example, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events).
   * Significant, uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation, ventricular fibrillation, or ventricular tachycardia).
   * Use of rate control drugs for arrhythmias (including beta blockers [such as metoprolol],acetylcholine, digoxin, and non-dihydropyridine calcium channel blockers diltiazem and verapamil).
   * Placement of a pacemaker for control of cardiac rhythm.
   * Requirement for inotropic support (including digoxin).
   * New York Heart Association (NYHA) Class II to IV heart failure.
   * Any other cardiac condition that in the opinion of the investigator could pose an additional risk for the participation in the study (example, pericardial effusion or restrictive cardiomyopathy).
   * Baseline prolongation of the rate-corrected QT interval (QTc; example, repeated demonstration of QTc interval >480 millisecond (msec), or history of congenital, long QT syndrome, or torsades de pointes).
7. With any of the following blood pressure conditions:

   * History of orthostatic hypotension or syncope that required medical intervention. Orthostatic hypotension is defined as a 20 millimeter of mercury (mmHg) fall in systolic blood pressure and/or a 10 mmHg fall in diastolic blood pressure within 2 to 5 minutes of quiet standing immediately after a 5-minute period of supine rest.
   * Postural orthostatic tachycardia syndrome (POTS) or postural tachycardia syndrome (defined as an increase in heart rate of >30 beats per minute over baseline after 10 minutes of quiet standing).
   * Hypertension that is unstable or not controlled by medication.
8. Seizures requiring antiepileptic treatment.
9. History of uncontrolled brain metastasis unless:

   * Previously treated with surgery, whole-brain radiation, or stereotactic radiosurgery.
   * Stable disease for ≥60 days, without steroid use (or stable steroid dose established for ≥28 days before the first dose of TAK-931).
10. Symptomatic and/or progressive central nervous system (CNS) metastases.
11. Ongoing medical conditions, such as acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before receiving the first dose of study drug.
12. Known history of human immunodeficiency virus (HIV) infection.
13. Known hepatitis B (HBV) surface antigen seropositive or detectable hepatitis C (HCV) infection viral load. Note: Participants who have positive hepatitis B core antibody or hepatitis B surface antibody can be enrolled but must have an undetectable hepatitis B viral load. Participants who have positive hepatitis C antibody must have an undetectable hepatitis C viral load.
14. Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption of study drug, such as total gastrectomy or GI conditions that could substantially modify gastric pH.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Kashiwa, Chiba
  - Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Kuboki Y, Shimizu T, Yonemori K, Kojima T, Kondo S, Koganemaru S, Iwasa S, Harano K, Koyama T, Lu V, Zhou X, Niu H, Yanai T, Garcia-Ribas I, Doi T, Yamamoto N. Safety, Tolerability, and Pharmacokinetics of TAK-931, a Cell Division Cycle 7 Inhibitor, in Patients with Advanced Solid Tumors: A Phase I First-in-Human Study. Cancer Res Commun. 2022 Nov 14;2(11):1426-1435. doi: 10.1158/2767-9764.CRC-22-0277. eCollection 2022 Nov. PMID 36970056
- [Derived] Martin JC, Sims JR, Gupta A, Bakin AV, Ohm JE. WEE1 inhibition augments CDC7 (DDK) inhibitor-induced cell death in Ewing sarcoma by forcing premature mitotic entry and mitotic catastrophe. Cancer Res Commun. 2022 Jun;2(6):471-482. doi: 10.1158/2767-9764.crc-22-0130. Epub 2022 Jun 20. PMID 36338546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 24 March 2016 to 21 December 2019.
Pre-assignment Details: Participants with advanced nonhematological solid tumors were enrolled to receive TAK-931 in 1 of the 4 treatment schedules: Schedule A, Schedule B, Schedule D and Schedule E. Schedules C and F were not conducted due to business reasons.
Groups:
- Schedule A: TAK-931 30 mg: TAK-931 30 milligram (mg), capsule, orally, once daily (QD) for 14 days in a 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule A: TAK-931 40 mg: TAK-931 40 mg, capsule, orally, once daily for 14 days in a 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule A: TAK-931 50 mg: TAK-931 50 mg, capsule, orally, once daily for 14 days in a 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule A: TAK-931 60 mg: TAK-931 60 mg, capsule, orally, once daily for 14 days in a 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule B: TAK-931 60 mg: TAK-931 60 mg, capsule, orally, once daily or twice daily (BID) for 7 days, followed by 7 days of rest and repeated (7 days on and 7 days off treatment) in each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule B: TAK-931 80 mg: TAK-931 80 mg, capsule, orally, once daily or twice daily for 7 days, followed by 7 days of rest and repeated (7 days on and 7 days off treatment) in each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule B: TAK-931 100 mg: TAK-931 100 mg, capsule, orally, once daily or twice daily for 7 days, followed by 7 days of rest and repeated (7 days on and 7 days off treatment) in each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule B: TAK-931 120 mg: TAK-931 120 mg, capsule, orally, once daily or twice daily for 7 days, followed by 7 days of rest and repeated (7 days on and 7 days off treatment) in each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule D: TAK-931 20 mg: TAK-931 20 mg, capsule, orally, once daily in each 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule D: TAK-931 30 mg: TAK-931 30 mg, capsule, orally, once daily in each 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule D: TAK-931 40 mg: TAK-931 40 mg, capsule, orally, once daily in each 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule E: TAK-931 100 mg: TAK-931 100 mg, capsule, orally, once daily on Days 1 and 2 followed by 5 days of rest and repeated weekly (2 days on and 5 days off treatment) in each 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule E: TAK-931 120 mg: TAK-931 120 mg, capsule, orally, once daily on Days 1 and 2 followed by 5 days of rest and repeated weekly (2 days on and 5 days off treatment) in each 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule E: TAK-931 150 mg: TAK-931 150 mg, capsule, orally, once daily on Days 1 and 2 followed by 5 days of rest and repeated weekly (2 days on and 5 days off treatment) in each 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
Period: Overall Study
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Started | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 3 | 14 | 3 | 3 | 7 | 5 | 5 | 6 | 6 | 5 | 4 | 3 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants who received any amount of study drug.
Groups:
- Schedule A: TAK-931 30 mg: TAK-931 30 mg, capsule, orally, once daily for 14 days in a 21-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Schedule B: TAK-931 60 mg: TAK-931 60 mg, capsule, orally, once daily or twice daily for 7 days, followed by 7 days of rest and repeated (7 days on and 7 days off treatment) in each 28-day treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent, death, or termination of the study by the sponsor.
- Total: Total of all reporting groups
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg | Total
Number analyzed (Participants) | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.81) | 56.7 (2.52) | 57.4 (11.99) | 59.3 (1.53) | 61.7 (3.21) | 52.4 (13.45) | 50.0 (8.15) | 59.8 (12.01) | 59.3 (6.56) | 62.7 (8.09) | 58.3 (17.41) | 59.5 (2.38) | 60.7 (13.58) | 62.8 (12.40) | 58.1 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 5 | 3 | 1 | 5 | 1 | 2 | 3 | 3 | 2 | 2 | 2 | 1 | 32
  Male | 3 | 1 | 11 | 0 | 2 | 4 | 5 | 4 | 3 | 3 | 4 | 2 | 1 | 5 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6 | 80
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 169.67 (8.663) | 159.70 (7.076) | 165.39 (6.727) | 155.03 (4.306) | 162.80 (11.012) | 163.64 (9.107) | 168.73 (7.387) | 167.40 (9.586) | 160.08 (12.071) | 156.43 (8.913) | 163.87 (7.469) | 162.43 (9.280) | 155.90 (12.612) | 165.92 (8.817) | 163.41 (8.890)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 70.07 (18.269) | 55.33 (3.099) | 62.06 (10.535) | 50.53 (3.707) | 58.03 (8.686) | 66.51 (16.750) | 71.00 (10.769) | 65.85 (10.783) | 59.63 (16.675) | 51.08 (10.167) | 56.25 (13.248) | 61.30 (13.851) | 53.27 (13.250) | 58.55 (13.772) | 60.91 (12.964)
Body Surface Area (BSA) [Median (Standard Deviation); unit: square meter (m˄2)] | 1.810 (0.2805) | 1.563 (0.0757) | 1.684 (0.1513) | 1.473 (0.0569) | 1.617 (0.1620) | 1.732 (0.2538) | 1.820 (0.1510) | 1.747 (0.1904) | 1.620 (0.2922) | 1.485 (0.1660) | 1.595 (0.2134) | 1.658 (0.2323) | 1.513 (0.2501) | 1.637 (0.2284) | 1.656 (0.2095)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Assessed by National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) Version 4.03
Description: Toxicity was evaluated by NCI CTCAE v4.03. DLT:any of following occurred events during Cycle 1 considered by investigator to be possibly related to therapy:1)Grade4 neutropenia,2)Febrile neutropenia lasting greater(>)1 hour,3)Grade greater than or equal to (>=)3 neutropenia with infection,4)Grade >=3 thrombocytopenia with bleeding,4)Grade 4 thrombocytopenia,5)delay in initiation of Cycle 2 by >14 days,6)Grade 2:<Grade 2 ejection fraction,7)other Grade 2 nonhematologic toxicities considered by investigator related to study drug and DLTs,8)who received <50 percent of doses of planned TAK-931 dosing in Cycle 1 for related AEs:<7 QD/<14 BID doses (Schedules A,B);<11 QD/<21 BID doses(Schedule D),<3 QD/<6 BID doses for(Schedule E),9)Grade >=3 nonhematologic toxicity except arthralgia/myalgia and fatigue, isolated >=Grade 3 laboratory abnormalities if it is asymptomatic and resolves to <=Grade 1 or baseline levels in <=7 days;inadequately treated Grade 3 nausea and/or vomiting and diarrhea.
Time Frame: Baseline up to Cycle 1 (Cycle length= 21 days [Schedules A, D and E] and 28 days [Schedule B])
Population: The DLT-evaluable population was defined as all participants who received at least 75% of their planned TAK-931 doses for their first cycle of treatment (unless interrupted by study drug-related AEs) and who had sufficient follow-up data to allow the investigators and sponsor to determine whether DLT occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
Participants | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2

2. Primary Outcome: Number of Participants With Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 30 days after the last dose of study drug or before initiation of new anti-cancer therapy (up to Day 499)
Population: The safety population was defined as all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
Participants | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 5 | 6 | 6 | 4 | 3 | 6

3. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration After First Dose of TAK-931
Time Frame: Cycle 1 Day 1: pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose (Cycle length= 21 days [Schedules A, D and E] and 28 days [Schedule B])
Population: The pharmacokinetic (PK) population was defined as all participants for whom there were sufficient dosing and TAK-931 concentration-time data to reliably estimate the PK parameter(s). Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 15 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
nanogram per milliliter (ng/mL) | 133 (22.6) | 229 (14.3) | 214 (40.9) | 265 (9.8) | 277 (19.0) | 302 (31.7) | 402 (24.5) | 454 (49.2) | 98.3 (37.0) | 149 (39.8) | 197 (31.5) | 462 (36.1) | 514 (15.9) | 499 (23.3)

4. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) After First Dose of TAK-931
Time Frame: as for outcome 3
Population: The PK population was defined as all participants for whom there were sufficient dosing and TAK-931 concentration-time data to reliably estimate the PK parameter(s). Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Median (Full Range); unit: hours
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 15 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
hours | 0.97 [0.93 to 1.93] | 1.05 [0.97 to 2.30] | 1.93 [0.45 to 2.13] | 3.88 [2.08 to 4.12] | 1.00 [0.42 to 1.03] | 4.00 [1.00 to 4.20] | 1.36 [0.47 to 3.98] | 1.05 [0.45 to 4.02] | 1.00 [0.93 to 2.17] | 2.13 [0.47 to 2.15] | 1.92 [0.87 to 3.95] | 2.00 [1.05 to 2.07] | 3.82 [1.88 to 4.05] | 2.07 [1.97 to 4.10]

5. Secondary Outcome: AUC24: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours After First Dose of TAK-931
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 15 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
hour*nanogram per milliliter (h*ng/mL) | 737 (24.1) | 1250 (14.6) | 1240 (31.8) | 2000 (33.8) | 1470 (17.9) | 2140 (35.9) | 2240 (23.9) | 2740 (29.5) | 494 (52.5) | 801 (32.3) | 1100 (28.2) | 2720 (20.0) | 3760 (48.9) | 3870 (35.9)

6. Secondary Outcome: AUC12: Area Under the Plasma Concentration-time Curve From 0 to 12 Hours After Multiple Doses of TAK-931
Time Frame: Cycle 1 Day 1: pre-dose and 0.5, 1, 2, 4, 6, 8 and 12 hours post-dose (Cycle length= 21 days [Schedules A, D and E] and 28 days [Schedule B])
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 15 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
h*ng/mL | 641 (22.2) | 1110 (13.4) | 1070 (29.9) | 1670 (30.5) | 1270 (12.2) | 1800 (32.8) | 1970 (23.2) | 2360 (28.8) | 431 (49.9) | 693 (30.3) | 956 (27.0) | 2280 (23.8) | 3110 (42.8) | 3160 (30.3)

7. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration After First Dose of TAK-931
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 15 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
h*ng/mL | 742 (24.3) | 1250 (14.7) | 1250 (32.0) | 2010 (34.0) | 1480 (17.7) | 2160 (36.0) | 2240 (23.7) | 2750 (29.5) | 491 (53.3) | 805 (32.4) | 1100 (28.2) | 2730 (20.5) | 3770 (49.3) | 3880 (35.8)

8. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration After Multiple Doses of TAK-931
Time Frame: Cycle 1 Day 8 (Schedule A and D), Cycle 1 Day 7 (Schedule B), Cycle 1 Day 9 (Schedule E): pre-dose and 0.5, 1, 2, 4, 6, 8, 12, and 24 hours post-dose (Cycle length= 21 days [Schedules A, D and E] and 28 days [Schedule B])
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 15 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
ng/mL | 133 (21.8) | 239 (16.2) | 231 (28.7) | 330 (23.9) | 218 (4.4) | 341 (54.0) | 380 (15.6) | 671 (73.6) | 104 (53.4) | 160 (34.1) | 193 (20.7) | 532 (39.9) | 654 (40.7) | 917 (22.1)

9. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) After Multiple Doses of TAK-931
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 8 | 6 | 6 | 6 | 6 | 5 | 4 | 3 | 6
hours | 2.02 [0.43 to 2.07] | 1.00 [0.93 to 1.90] | 1.91 [0.95 to 3.88] | 1.95 [0.92 to 2.08] | 2.00 [0.50 to 2.17] | 2.01 [0.90 to 3.90] | 1.90 [1.00 to 4.12] | 1.92 [0.98 to 4.12] | 1.50 [0.97 to 2.02] | 2.00 [0.9 to 3.97] | 1.08 [0.92 to 2.13] | 1.49 [0.95 to 4.07] | 2.07 [1.9 to 2.18] | 2.08 [0.92 to 2.20]

10. Secondary Outcome: AUC24: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours After Multiple Doses of TAK-931
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 8 | 6 | 6 | 6 | 6 | 5 | 4 | 3 | 6
h*ng/mL | 799 (19.3) | 1400 (15.4) | 1320 (33.6) | 2210 (30.5) | 1650 (10.4) | 2220 (39.8) | 2620 (26.8) | 4410 (81.8) | 600 (49.1) | 958 (46.1) | 1140 (41.2) | 3760 (28.6) | 4830 (55.6) | 6260 (32.2)

11. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration After Multiple Doses of TAK-931
Time Frame: as for outcome 8
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 8 | 6 | 6 | 6 | 6 | 5 | 4 | 3 | 6
h*ng/mL | 805 (19.4) | 1410 (15.0) | 1330 (33.9) | 2220 (30.8) | 1650 (10.4) | 2230 (39.8) | 2630 (27.4) | 4420 (81.0) | 603 (49.2) | 964 (46.4) | 1150 (41.3) | 3770 (28.7) | 4840 (55.8) | 6280 (32.2)

12. Secondary Outcome: Schedule A, B and D: Change From Baseline in Phosphorylated Minichromosome Maintenance Complex-2 (pMCM2) (Ser40) Levels in Skin Based on Histological Score Nuclei (H-score) After Multiple Doses Of TAK-931
Description: H-score were a composite score that comprised of intensity and percentage of staining and were used for assessing amount of protein (in this case pMCM2 [Ser40]) present in a tissue sample. The composite score obtained by H-score is derived by adding of the percentages of cell staining at each intensity level multiplied by the weighted intensity of staining (0 [no staining], 1+ [weak staining], 2+ [medium staining], 3+ [strong staining]). The H-score has a range of 0 to 300. Lower H-scores represent lower expression of pMCM2 (Ser40) in the tissue sample, while higher scores represent stronger expression of pMCM2 (Ser40) in the tissue samples.
Time Frame: Cycle 1 Day 1 pre-dose up to any dosing day after 3 consecutive days post-dose (up to Cycle 1 Day 8 [Schedule A and D]; Cycle 1 Day 7 [Schedule B]; Cycle 1 Day 12 [Schedule D]) (Cycle Length of Schedules A and D = 21 days; and Schedule B= 28 days)
Population: Pharmacodynamics population: all participants who received at least the first dose of TAK-931, had a baseline skin punch biopsy sample, and had at least 1 additional postbaseline skin punch biopsy sample. Overall number analyzed "N": participants who were evaluable for the outcome measure. Number analyzed "n": participants who were evaluable for this outcome measure for given categories. Data for this outcome measure was not collected and analyzed for Schedule E Cohorts due to business reasons.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg
Number analyzed (Participants) | 3 | 3 | 16 | 3 | 3 | 9 | 0 | 0 | 6 | 6 | 0
score on a scale
  Baseline: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 5 | 0 | 0 | 6 | 3 | 0
  Baseline | 18.467 (8.4506) | 19.533 (3.7754) | 10.500 (5.8477) | 10.933 (1.9425) | 4.400 (2.9597) | 12.720 (2.0229) |  |  | 22.050 (24.5239) | 33.317 (23.4266) |
  Schedule B: Change at Cycle 1 Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 0
  Schedule B: Change at Cycle 1 Day 7 |  |  |  |  | -3.733 (3.1770) | -9.180 (7.2589) |  |  |  |  |
  Schedule A and D: Change at Cycle 1 Day 8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 0 | 0 | 0 | 0 | 4 | 3 | 0
  Schedule A and D: Change at Cycle 1 Day 8 | -7.533 (2.9280) | -6.667 (10.5078) | -6.743 (8.7444) | -9.933 (2.2030) |  |  |  |  | -5.900 (4.2379) | -26.883 (24.5978) |
  Schedule D: Change at Cycle 1 Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Schedule D: Change at Cycle 1 Day 12 |  |  |  |  |  |  |  |  | -67.100 |  |

13. Secondary Outcome: Schedule A, B and D: Change From Baseline in pMCM2 (Ser40) Levels in Skin Based on Positive Index After Multiple Doses Of TAK-931
Description: Positive index was calculated by taking the number of cells staining positive for the marker over the total number of cells.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of cell
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg
Number analyzed (Participants) | 3 | 3 | 16 | 3 | 3 | 9 | 0 | 0 | 6 | 6 | 0
percentage of cell
  Baseline: number analyzed (Participants) | 3 | 3 | 14 | 3 | 3 | 5 | 0 | 0 | 6 | 3 | 0
  Baseline | 0.08600 (0.039950) | 0.08533 (0.019425) | 0.04429 (0.021780) | 0.04800 (0.006928) | 0.02000 (0.013856) | 0.05080 (0.007694) |  |  | 0.10217 (0.126757) | 0.15200 (0.128829) |
  Schedule B: Change at Cycle 1 Day 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 0
  Schedule B: Change at Cycle 1 Day 7 |  |  |  |  | -0.01667 (0.015144) | -0.01916 (0.063995) |  |  |  |  |
  Schedule A and D: Change at Cycle 1 Day 8: number analyzed (Participants) | 3 | 3 | 14 | 3 | 0 | 0 | 0 | 0 | 4 | 3 | 0
  Schedule A and D: Change at Cycle 1 Day 8 | -0.03037 (0.014191) | -0.02386 (0.046889) | -0.02643 (0.033014) | -0.04125 (0.008245) |  |  |  |  | -0.02150 (0.018930) | -0.12436 (0.134410) |
  Schedule D: Change at Cycle 1 Day 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Schedule D: Change at Cycle 1 Day 12 |  |  |  |  |  |  |  |  | -0.33900 |  |

14. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as percentage of participants who had achieved complete response (CR) and partial response (PR), as measured by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST V 1.1). CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR: was at least a 30 percent (%) decrease in sum of diameter (SOD) of target lesions, taking as reference the baseline SOD.
Time Frame: From date of first dose to the date of first documentation of progressive disease (PD) or death due to any cause, which ever occurred first (up to Month 45)
Population: The response-evaluable population is defined as participants who receive at least 1 dose of study drug, have measurable disease at baseline, and at least 1 post-baseline response assessment. Here "overall number of participants analyzed" are participants who were available for this outcome measure assessment at given time period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 15 | 3 | 3 | 8 | 6 | 6 | 6 | 5 | 6 | 3 | 3 | 5
percentage of participants | 33 [1 to 91] | 0 [0 to 71] | 7 [0 to 32] | 33 [1 to 91] | 0 [0 to 71] | 0 [0 to 37] | 17 [0 to 64] | 17 [0 to 64] | 0 [0 to 46] | 0 [0 to 52] | 0 [0 to 46] | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 52]

15. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of first dose to the date of first documentation of PD or death due to any cause, whichever occurs first, as measured by RECIST V1.1. PD: 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PFS was analyzed using the Kaplan-Meier method.
Time Frame: From date of first dose to the date of first documentation of PD or death due to any cause, which ever occurred first (up to Month 45)
Population: The safety population was defined as all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 3 | 3 | 16 | 3 | 3 | 9 | 6 | 6 | 6 | 6 | 6 | 4 | 3 | 6
months | 4.2 [1.74 to 9.20] | 2.1 [0.53 to 3.29] | 2.0 [1.68 to 5.32] | 4.8 [3.32 to 6.34] | 3.1 [0.92 to 5.85] | 2.8 [1.58 to 3.25] | 2.1 [0.79 to 6.21] | 4.2 [1.84 to 6.64] | 1.9 [1.41 to 2.10] | 3.9 [1.91 to 8.05] | 2.1 [1.18 to 15.24] | 1.9 [0.39 to 3.91] | 1.9 [1.05 to 4.37] | 2.6 [0.53 to 5.88]

16. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time from the date of first documentation of a response (CR or PR) to the date of first documentation of PD, as measured by RECIST V 1.1. CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: was at least a 30% decrease in SOD of target lesions, taking as reference the baseline SOD. PD: 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. DOR was analyzed using the Kaplan-Meier method.
Time Frame: From the date of first documentation of response to the date of first documentation of PD (up to Month 45)
Population: The response-evaluable population is defined as participants who receive at least 1 dose of study drug, have measurable disease at baseline, and at least 1 post-baseline response assessment. Responders without documentation of PD were censored at the date of last response assessment that is stable disease or better.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
months | 2.1 |  | 2.7 | 2.2 |  |  | 4.2 | 0.0 |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events (AEs) that started after the first dose of study drug through 30 days after the last dose of study drug or before initiation of new anti-cancer therapy (whichever occurred first) (up to Day 499)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Schedule A: TAK-931 30 mg | Schedule A: TAK-931 40 mg | Schedule A: TAK-931 50 mg | Schedule A: TAK-931 60 mg | Schedule B: TAK-931 60 mg | Schedule B: TAK-931 80 mg | Schedule B: TAK-931 100 mg | Schedule B: TAK-931 120 mg | Schedule D: TAK-931 20 mg | Schedule D: TAK-931 30 mg | Schedule D: TAK-931 40 mg | Schedule E: TAK-931 100 mg | Schedule E: TAK-931 120 mg | Schedule E: TAK-931 150 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/16 | 0/3 | 0/3 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 5/16 | 2/3 | 1/3 | 2/9 | 1/6 | 1/6 | 1/6 | 1/6 | 3/6 | 2/4 | 0/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 16/16 | 3/3 | 3/3 | 9/9 | 6/6 | 6/6 | 5/6 | 6/6 | 6/6 | 4/4 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A: TAK-931 30 mg (N=3) | Schedule A: TAK-931 40 mg (N=3) | Schedule A: TAK-931 50 mg (N=16) | Schedule A: TAK-931 60 mg (N=3) | Schedule B: TAK-931 60 mg (N=3) | Schedule B: TAK-931 80 mg (N=9) | Schedule B: TAK-931 100 mg (N=6) | Schedule B: TAK-931 120 mg (N=6) | Schedule D: TAK-931 20 mg (N=6) | Schedule D: TAK-931 30 mg (N=6) | Schedule D: TAK-931 40 mg (N=6) | Schedule E: TAK-931 100 mg (N=4) | Schedule E: TAK-931 120 mg (N=3) | Schedule E: TAK-931 150 mg (N=6)
Oncologic complications and emergencies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mediastinal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to specified sites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatic neoplasms malignant (excl islet cell and carcinoid) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenias 0 1 (33) 0 1 (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stenosis and obstruction NEC (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal and small intestinal stenosis and obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal inflammatory disorders NEC (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea and vomiting symptoms (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis, bacteraemia, viraemia and fungaemia NEC (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal and gastrointestinal infections (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract and lung infections (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appetite disorders (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Central nervous system haemorrhages and cerebrovascular accidents (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased intracranial pressure disorders (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizures and seizure disorders NEC (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract inflammatory and immunologic conditions (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenic conditions (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary abnormalities (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A: TAK-931 30 mg (N=3) | Schedule A: TAK-931 40 mg (N=3) | Schedule A: TAK-931 50 mg (N=16) | Schedule A: TAK-931 60 mg (N=3) | Schedule B: TAK-931 60 mg (N=3) | Schedule B: TAK-931 80 mg (N=9) | Schedule B: TAK-931 100 mg (N=6) | Schedule B: TAK-931 120 mg (N=6) | Schedule D: TAK-931 20 mg (N=6) | Schedule D: TAK-931 30 mg (N=6) | Schedule D: TAK-931 40 mg (N=6) | Schedule E: TAK-931 100 mg (N=4) | Schedule E: TAK-931 120 mg (N=3) | Schedule E: TAK-931 150 mg (N=6)
Nausea (Gastrointestinal disorders) | 0 | 2 | 10 | 3 | 1 | 9 | 5 | 6 | 0 | 3 | 2 | 1 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 8 | 2 | 1 | 7 | 5 | 6 | 1 | 2 | 3 | 1 | 2 | 5
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 2 | 0 | 7 | 2 | 4 | 0 | 0 | 2 | 1 | 2 | 4
White blood cell count decreased (Investigations) | 1 | 0 | 6 | 1 | 0 | 1 | 0 | 4 | 1 | 3 | 3 | 1 | 1 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 2 | 1 | 5 | 3 | 4 | 0 | 1 | 2 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 0 | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 1 | 5 | 5 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Cardiac disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Application site pruritus (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vagus nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02699749/SAP_000.pdf
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT02699749/Prot_001.pdf